CLINICAL TRIAL: NCT06484036
Title: Effectiveness of Periodontitis Treatment on the Metabolic Activity of Symptomatic Carotid Atherosclerotic Plaque Responsible for Ischemic Stroke: a Multicenter Randomized Controlled Trial: a Multicenter Randomized Controlled Trial
Brief Title: Effectiveness of Periodontitis Treatment on the Metabolic Activity of Symptomatic Carotid Atherosclerotic Plaque Responsible for Ischemic Stroke
Acronym: PerioStroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP230861
Record Dates: First submitted 2024-06-24; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-05

CONDITIONS: Severe Periodontitis; Ischemic Stroke
Keywords: PET scan; Severe Periodontitis; Ischemic Stroke
MeSH Terms: conditions — Periodontitis; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: This is a multicenter, open-label, randomized controlled superiority trial in 2 parallel groups with adjudication of the primary endpoint blinded to the randomization group and centrally (PET reading).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with periodontal treatment strategy (Experimental): Group with periodontal treatment strategy, in addition to routine care and secondary prevention of ischemic stroke
  Interventions: Procedure: periodontal treatment strategy
- Group without periodontal treatment (No Intervention): Group without periodontal treatment, with routine care and secondary prevention of ischemic stroke

INTERVENTIONS:
Procedure: periodontal treatment strategy — Periodontal treatment sessions (Experimental Group only) (1 to 3 months) after randomization
  Arms: Group with periodontal treatment strategy

SUMMARY:
Cardiovascular disease is the world's leading cause of death. Atherothrombosis is a common cause of ischemic stroke.

A strong epidemiological link has been established between periodontitis and the risk of stroke. It shares common risk factors with atherothrombosis, and its severe form is associated with low-grade systemic inflammation and daily low-intensity bacteremia. Atherothrombosis is a frequent cause of ischemic stroke.

Periodontal bacteria have been found within atheromatous plaques, correlated with a greater risk of rupture.

Thus, periodontitis could be a modifiable risk factor for atherothrombosis and future vascular events: its early diagnosis and treatment could have a major impact on cardiovascular prevention.

Hypothesis: In patients with periodontitis who have had an ischemic stroke, periodontal treatment may reduce atherosclerotic plaque activity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Minor ischemic stroke of the anterior circulation (NIHSS ≤ 5) of atherothrombotic origin according to the TOAST scale <30 days
* Atheroma plaque of the ipsilateral carotid bulb >30% not eligible for intervention (endarterectomy or angioplasty-stenting)
* Severe periodontitis (stage 3 or 4)
* Signed informed consent
* Affiliation to a social security scheme

Exclusion Criteria:

* < 6 teeth
* Without independent oral hygiene
* Contraindications to PET scan
* Known allergy to fluoro-deoxyglucose and its excipient
* Immunosuppressive treatment
* Uncontrolled diabetes
* High risk of infective endocarditis
* Organ transplant pending
* Progressive infectious diseases
* Active smoking not stopped
* Patient deprived of liberty by judicial or administrative decision
* Patient under legal protection (guardianship, curatorship)
* Participation in another interventional research involving humans or being in the exclusion period following previous research involving humans
* Pregnant or breastfeeding woman Patient under AME (state medical aid)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Percentage evolution (relative evolution) of patients with Target-to-Background (TBR) becomes <1.6 (threshold). | At 6 months
  The evolution of the metabolic activity of the atherosclerotic plaque measured by the Target-to-Background ratio (TBR) measured by PET scan after injection of 18-FDG at 6 months versus at baseline in percentage evolution (relative evolution) and in number of patients for whom the TBR becomes <1.6 (threshold).
Number of patients with Target-to-Background (TBR) becomes <1.6 (threshold). | At 6 months
  The evolution of the metabolic activity of the atherosclerotic plaque measured by the Target-to-Background ratio (TBR) measured by PET scan after injection of 18-FDG at 6 months versus at baseline in percentage evolution (relative evolution) and in number of patients for whom the TBR becomes <1.6 (threshold).

SECONDARY OUTCOMES:
Absolute change on Target-to-Background (TBR) ratio | At 6 months
  Nominal change in atherosclerotic plaque metabolic activity measured by Target-to-Background (TBR) ratio measured by PET scan after 18-FDG injection at 6 months versus at baseline (absolute change).
Proportion of TBR success becomes <1.6 | At 6 months
cardiovascular event | At 12 months
ischemic stroke | At 12 months
Atherothrombotic event | At 12 months
Acute coronary syndrome | At 12 months
Limb ischemia | At 12 months
Mortality | At 12 months
Difference in hs-CRP measurement | 6 months and 12 months
Difference in Lp-PLA2 measurement | 6 months and 12 months
Serious and non-serious adverse events | up to 12 Months